CLINICAL TRIAL: NCT06588296
Title: Efficacy and Safety of Ixekizumab or Ixekizumab Concomitantly Administered With Tirzepatide in Adult Participants With Active Psoriatic Arthritis and Obesity or Overweight: A Phase 3b, Randomized, Multicenter, Open-Label Study (TOGETHER-PsA)
Brief Title: Ixekizumab Concomitantly Administered With Tirzepatide in Adults With Psoriatic Arthritis and Obesity or Overweight
Acronym: TOGETHER-PsA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27241; I1F-MC-RHDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis; Obesity
MeSH Terms: conditions — Arthritis, Psoriatic; Obesity | interventions — ixekizumab; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental): Ixekizumab administered subcutaneous (SC).
  Interventions: Drug: Ixekizumab
- Ixekizumab and Tirzepatide (Experimental): Ixekizumab concomitantly administered with tirzepatide SC.
  Interventions: Drug: Ixekizumab; Drug: Tirzepatide

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Ixekizumab and Tirzepatide

SUMMARY:
The main purpose of this study is to demonstrate that when participants with psoriatic arthritis and obesity or overweight in the presence of at least 1 weight-related comorbid condition receive ixekizumab and tirzepatide concomitantly administered, participants see improvement in their psoriatic arthritis and achieve weight reduction compared to when receiving ixekizumab.

Participation in this study includes up to 12 visits and could last up to 61 weeks including screening, open label treatment period, and post-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have signs and/or symptoms or documented diagnosis of Psoriatic Arthritis (PsA) for at least 6 months and currently fulfilling the classification of Psoriatic Arthritis (CASPAR) criteria.
* Have active PsA, defined as the presence of at least 3 of 68 tender joints and at least 3 of 66 swollen joints.
* Have obesity, body mass index of ≥30 kilograms per meter squared (BMI ≥30 kg/m²) or overweight (BMI ≥27 to <30 kg/m²) in the presence of at least 1 of these weight-related comorbid conditions (hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease, or T2DM).

Exclusion Criteria:

Medical Conditions

* Have Type 1 Diabetes Mellitus (T1DM).
* Have insulin-treated Type 2 Diabetes Mellitus (T2DM).
* Have a prior or planned surgical treatment for obesity.
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia (MEN) syndrome type 2.
* Have active, or a history of inflammatory bowel disease (Crohn's or ulcerative colitis).
* Have a diagnosis or history of malignant disease within the 5 years prior to randomization, with the following exceptions:

  * basal cell or squamous epithelial carcinomas of the skin that have been resected, with no evidence of metastatic disease for 3 years.
  * cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to randomization.
* Have a serious disorder or illness other than PsA.
* Have a history of chronic or acute pancreatitis.
* Have any prior use of ixekizumab or tirzepatide.
* Diagnosis of other inflammatory arthritis, such as Rheumatoid Arthritis (RA), ankylosing spondylitis, reactive arthritis, gout, or enteropathic arthritis.
* Have a previous failure or intolerance to an interleukin 17 inhibitor (IL-17i) or glucagon-like peptide 1 (GLP-1) receptor agonists.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Simultaneously Achieved American College of Rheumatology (ACR) ACR50 and at Least a 10% Weight Reduction | Baseline up to Week 36
  ACR50 is defined as at least 50% improvement in the ACR core set values. The percentage improvement in the ACR scores is determined by an improvement of at least 50% in the number of Tender Joint Count (TJC) (0-68) and Swollen Joint Count (SJC) (0-66) and an improvement of at least 50% in at least 3 of these 5 assessments:
  1. Patient's Assessment of Arthritis Pain Visual Analog Scale (VAS)
  2. Patient's Global Assessment of Disease Activity Numeric Rating Scale (PaGADA _NRS)
  3. Physician's Global Assessment of Disease Activity Numeric Rating Scale (PhGADA NRS)
  4. Patient's Assessment of Physical Function as measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) or
  5. Acute phase reactant as measured by High-Sensitivity C-Reactive Protein (hsCRP)

SECONDARY OUTCOMES:
Percentage of Participants Simultaneously Achieving American College of Rheumatology (ACR) ACR20 and at Least a 5% Weight Reduction | Baseline up to Week 36
  ACR20 is defined as at least 20% improvement in the ACR core set values. The percentage improvement in the ACR scores is determined by an improvement of at least 20% in the number of TJC (0-68) and SJC (0-66) and an improvement of at least 20% in at least 3 of these 5 assessments:
  1. Patient's Assessment of Arthritis Pain Visual Analog Scale (VAS)
  2. Patient's Global Assessment of Disease Activity Numeric Rating Scale (PaGADA _NRS)
  3. Physician's Global Assessment of Disease Activity Numeric Rating Scale (PhGADA NRS)
  4. Patient's Assessment of Physical Function as measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) or
  5. Acute phase reactant as measured by High-Sensitivity C-Reactive Protein (hsCRP)
Percentage of Participants Achieving ACR50 | Baseline up to Week 36
  ACR50 is defined as at least 50% improvement in the ACR core set values. The percentage improvement in the ACR scores is determined by an improvement of at least 50% in the number of TJC (0-68) and SJC (0-66) and an improvement of at least 50% in at least 3 of these 5 assessments:
  1. Patient's Assessment of Arthritis Pain Visual Analog Scale (VAS)
  2. Patient's Global Assessment of Disease Activity Numeric Rating Scale (PaGADA _NRS)
  3. Physician's Global Assessment of Disease Activity Numeric Rating Scale (PhGADA NRS)
  4. Patient's Assessment of Physical Function as measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI) or
  5. Acute phase reactant as measured by High-Sensitivity C-Reactive Protein (hsCRP)
Percentage of Participants Achieving at Least a 10% Weight Reduction | Baseline up to Week 36
  Percentage of Participants Who Achieved at Least a 10% Weight Reduction

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (86):
- United States (81):
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Chandler, Chandler, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Flagstaff, Flagstaff, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Gilbert, Gilbert, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Glendale, Glendale, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Mesa, Mesa, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Phoenix PV, Phoenix, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Sun City, Sun City, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson, Tucson, Arizona
  - AARA Clinical Research - Arizona Arthritis & Rheumatology Associates - Tucson Southeast, Tucson, Arizona
  - Medvin Clinical Research - Apple Valley, Apple Valley, California
  - Medvin Clinical Research - Covina, Covina, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - Purushotham & Akther Kotha MD, Inc, La Mesa, California
  - Medvin Clinical Research - Riverside, Riverside, California
  - Rheumatology Center of San Diego, San Diego, California
  - Medvin Clinical Research - Temecula, Temecula, California
  - Cohen Medical Centers, Thousand Oaks, California
  - Medvin Clinical Research - Tujunga, Tujunga, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - NeoClinical Research, Hialeah, Florida
  - South Florida Rheumatology, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Vida Clinical Research, Kissimmee, Florida
  - Life Clinical Trials, Margate, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Vitalia Medical Research, Palm Beach Gardens, Florida
  - Sarasota Arthritis Center, Sarasota, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - International Center for Research, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Southeastern Rheumatology Alliance dba Arthritis Center of North Georgia, Gainesville, Georgia
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - St. Luke's Clinic, Boise, Idaho
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Greater Chicago Specialty Physicians, Schaumburg, Illinois
  - Arnold Arthritis & Rheumatology, Skokie, Illinois
  - Willow Rheumatology and Wellness PLLC, Willowbrook, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Accurate Clinical Research, Inc, Lake Charles, Louisiana
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Advanced Rheumatology, PC, Okemos, Michigan
  - Saint Paul Rheumatology, Eagan, Minnesota
  - AARA Clinical Research - Kansas City Physician Partners - North, Kansas City, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Arthritis Consultants, Inc., St Louis, Missouri
  - Logan Health Research, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - St. Lawrence Health System, Canton, New York
  - Onsite Clinical Solutions, LLC - Brenner Ave, Salisbury, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - RAO Research LLC, Oklahoma City, Oklahoma
  - Essential Medical Research, Tulsa, Oklahoma
  - Summit Headlands, Portland, Oregon
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - AARA Clinical Research - Murfreesboro Medical Clinic, Murfreesboro, Tennessee
  - Tekton Research, LLC., Austin, Texas
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions - Colleyville, Colleyville, Texas
  - Arthritis Care of Texas, Corpus Christi, Texas
  - AARA Clinical Research - Lone Star Arthritis and Rheumatology Associates - Fort Worth, Fort Worth, Texas
  - Accurate Clinical Research, Inc, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - AARA Clinical Research - Lone Star Arthritis and Rheumatology Associates - Irving, Irving, Texas
  - Biopharma Informatic, LLC, Katy, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Valley Arthritis Center, McAllen, Texas
  - SouthWest Rheumatology Research, LLC, Mesquite, Texas
  - Advanced Rheumatology of Houston - Woodlands, The Woodlands, Texas
  - DM Clinical Research - TRA, Tomball, Texas
  - Overlake Arthritis and Osteoporosis Center, Bellevue, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
- Puerto Rico (5):
  - Centro Reumatologico Caguas, Caguas
  - Reuviva Research Center, Guaynabo
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - Caribbean Medical Research Center, San Juan
  - Mindful Medical Research, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/